CLINICAL TRIAL: NCT00970424
Title: A Phase III, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate the Safety and Efficacy of Dutogliptin in Patients With Type 2 Diabetes Mellitus on Background Treatment With Pioglitazone
Brief Title: Safety and Efficacy of Dutogliptin in Patients With Type 2 Diabetes Mellitus (T2DM) on Background Therapy With Pioglitazone
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Collaborators: Phenomix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DUT-MD-304
Record Dates: First submitted 2009-09-01; First posted 2009-09-02 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-09

CONDITIONS: Diabetes Mellitus, Type II
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dutogliptin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): placebo, oral tablet administered once daily on background of pioglitazone
  Interventions: Drug: Placebo
- 2 (Experimental): dutogliptin, oral tablet administered once daily on background of pioglitazone
  Interventions: Drug: Dutogliptin

INTERVENTIONS:
Drug: Placebo — placebo, oral tablet administered once daily on background of pioglitazone
  Arms: 1
Drug: Dutogliptin — dutogliptin, oral tablet administered once daily on background of pioglitazone
  Arms: 2

SUMMARY:
This study will evaluate the safety and efficacy of dutogliptin in patients with type 2 diabetes mellitus (T2DM) who are receiving background treatment with pioglitazone.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus, diagnosed at least 3 months prior to Screening (Visit 1)
* BMI 20 to 48 kg/m2, inclusive
* HbA1c 7.0% - 10.0%, inclusive
* Age 18 to 85 years, inclusive

Exclusion Criteria:

* Currently taking more than one oral hypoglycemic agent
* Type 1 diabetes mellitus

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 252 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1c Level (HbA1c) | HbA1c is drawn at Visit 1 (Week -16 to -4), Visit 3 (Week -2), Visit 4 (Week 0), Visit 5 (Week 4), Visit 6 (Week 10), Visit 7 (Week 18) and Week 8 (Week 26)

SECONDARY OUTCOMES:
Fasting Plasma Glucose Level (FPG) | FPG is drawn at Visit 1 (Week -16 to -4), Visit 2 (Week -4), Visit 3 (Week -2), Visit 4 (Week 0), Visit 5 (Week 4), Visit 6 (Week 10), Visit 7 (Week 18) and Visit 8 (Week 26).

CONTACTS AND LOCATIONS:
Overall Officials: Kaity Posada, PharmD, Study Director — Forest Research Institute, a subsidiary of Forest Laboratories, Inc.
Locations (118):
- United States (89):
  - Forest Investigative Site 064, Birmingham, Alabama
  - Forest Investigative Site 020, Birmingham, Alabama
  - Forest Investigative Site 059, Chandler, Arizona
  - Forest Investigative Site 096, Litchfield, Arizona
  - Forest Investigative Site 098, Phoenix, Arizona
  - Forest Investigative Site 044, Scottsdale, Arizona
  - Forest Investigative Site 087, Tucson, Arizona
  - Forest Investigative Site 061, Anaheim, California
  - Forest Investigative Site 041, Chula Vista, California
  - Forest Investigative Site 049, Encinitas, California
  - Forest Investigative Site 022, Greenbrae, California
  - Forest Investigative Site 047, Harbor City, California
  - Forest Investigative Site 010, Huntington Park, California
  - Forest Investigative Site 111, Northridge, California
  - Forest Investigative Site 031, Riverside, California
  - Forest Investigative Site 091, Roseville, California
  - Forest Investigative Site 067, Sacramento, California
  - Forest Investigative Site 112, Santa Ana, California
  - Forest Investigative Site 011, Walnut Creek, California
  - Forest Investigative Site 063, West Hills, California
  - Forest Investigative Site 115, Colorado Springs, Colorado
  - Forest Investigative Site 073, Clearwater, Florida
  - Forest Investigative Site 004, Daytona Beach, Florida
  - Forest Investigative Site 052, DeLand, Florida
  - Forest Investigative Site 062, Jacksonville, Florida
  - Forest Investigative Site 021, Miami, Florida
  - Forest Investigative Site 050, Miami, Florida
  - Forest Investigative Site 122, Miami, Florida
  - Forest Investigative Site 015, Orlando, Florida
  - Forest Investigative Site 018, Sarasota, Florida
  - Forest Investigative Site 075, St. Petersburg, Florida
  - Forest Investigative Site 026, West Palm Beach, Florida
  - Forest Investigative Site 045, Atlanta, Georgia
  - Forest Investigative Site 079, Augusta, Georgia
  - Forest Investigative Site 009, Meridian, Idaho
  - Forest Investigative Site 60, Melrose Park, Illinois
  - Forest Investigative Site 030, Peoria, Illinois
  - Forest Investigative Site 100, Evansville, Indiana
  - Forest Investigative Site 097, Evansville, Indiana
  - Forest Investigative Site 053, Kansas City, Kansas
  - Forest Investigative Site 008, Wichita, Kansas
  - Forest Investigative Site 078, Erlanger, Kentucky
  - Forest Investigative Site 024, Madisonville, Kentucky
  - Forest Investigative Site 034, Covington, Louisiana
  - Forest Investigative Site 035, Baltimore, Maryland
  - Forest Investigative Site 046, Oxon Hill, Maryland
  - Forest Investigative Site 118, New Bedford, Massachusetts
  - Forest Investigative Site 007, Waltham, Massachusetts
  - Forest Investigative Site 002, Dearborn, Michigan
  - Forest Investigative Site 029, Saint Clair Shores, Michigan
  - Forest Investigative Site 054, Edina, Minnesota
  - Forest Investigative Site 013, Grand Island, Nebraska
  - Forest Investigative Site 072, Las Vegas, Nevada
  - Forest Investigative Site 065, Las Vegas, Nevada
  - Forest Investigative Site 081, New Hyde Park, New York
  - Forest Investigative Site 016, New York, New York
  - Forest Investigative Site 094, Charlotte, North Carolina
  - Forest Investigative Site 051, Charlotte, North Carolina
  - Forest Investigative Site 117, Charlotte, North Carolina
  - Forest Investigative Site 058, Lenoir, North Carolina
  - Forest Investigative Site 038, Morehead City, North Carolina
  - Forest Investigative Site 040, Salisbury, North Carolina
  - Forest Investigative Site 039, Akron, Ohio
  - Forest Investigative Site 023, Cincinnati, Ohio
  - Forest Investigative Site 043, Columbus, Ohio
  - Forest Investigative Site 057, Dayton, Ohio
  - Forest Investigative Site 032, Kettering, Ohio
  - Forest Investigative Site 149, Norman, Oklahoma
  - Forest Investigative Site 102, Ashland, Oregon
  - Forest Investigative Site 005, Eugene, Oregon
  - Forest Investigative Site 037, Harleysville, Pennsylvania
  - Forest Investigative Site 066, Philadelphia, Pennsylvania
  - Forest Investigative Site 036, Tipton, Pennsylvania
  - Forest Investigative Site 103, Greer, South Carolina
  - Forest Investigative Site 090, Manning, South Carolina
  - Forest Investigative Site 033, Pelzer, South Carolina
  - Forest Investigative Site 114, Chattanooga, Tennessee
  - Forest Investigative Site 104, Chattanooga, Tennessee
  - Forest Investigative Site 099, Arlington, Texas
  - Forest Investigative Site 056, Corpus Christi, Texas
  - Forest Investigative Site 017, Dallas, Texas
  - Forest Investigative Site 124, Dallas, Texas
  - Forest Investigative Site 106, Houston, Texas
  - Forest Investigative Site 014, Irving, Texas
  - Forest Investigative Site 109, San Antonio, Texas
  - Forest Investigative Site 076, Salt Lake City, Utah
  - Forest Investigative Site 028, Virginia Beach, Virginia
  - Forest Investigative Site 092, Spokane, Washington
  - Forest Investigative Site 027, Milwaukee, Wisconsin
- Forest Investigative Site 209, Mogilev, Belarus, Belarus
- Germany (3):
  - Forest Investigative Site 401, Dresden, Germany
  - Forest Investigative Site 402, Dresden, Germany
  - Forest Investigative Site 403, Mainz, Germany
- India (14):
  - Forest Investigative Site 614, Vijayawada, Andhra Pradesh
  - Forest Investigative Site 618, Ahmedabad, Gujarat
  - Forest Investigative Site 620, Haryāna, Karnal
  - Forest Investigative Site 607, Bangalore, Karnataka
  - Forest Investigative Site 606, Bangalore, Karnataka
  - Forest Investigative Site 602, Bangalore, Karnataka
  - Forest Investigative Site 604, Bangalore, Karnataka
  - Forest Investigative Site 601, Mangalore, Karnataka
  - Forest Investigative Site 616, Nagpur, Maharashtra
  - Forest Investigative Site 617, Nashik, Maharashtra
  - Forest Investigative Site 612, Pune, Maharashtra
  - Forest Investigative Site 603, Channi, Tamil Nadu
  - Forest Investigative Site 613, Chennai, Tamil Nadu
  - Forest Investigative Site 615, Vellore, Tamil Nadu
- Lithuania (4):
  - Forest Investigative Site 702, Kaunas, Lithunia
  - Forest Investigative Site 703, Kaunas, Lithunia
  - Forest Investigative Site 704, Klaipėda, Lithunia
  - Forest Investigative Site 705, Vilnius, Lithunia
- Romania (7):
  - Forest Investigative Site 909, Bacau, Romania
  - Forest Investigative Site 906, Bucharest, Romania
  - Forest Investigative Site 908, Bucharest, Romania
  - Forest Investigative Site 903, Satu Mare, Romania
  - Forest Investigative Site 901, Sibiu, Romania
  - Forest Investigative Site 905 Romania, Tg Mures, Romania
  - Forest Investigative Site 902, Timișoara, Romania